CLINICAL TRIAL: NCT01729338
Title: Phase II Subcutaneous VELCADE and Oral Cyclophosphamide-based Induction + Sequential VELCADE and Revlimid Maintenance for Newly Diagnosed Multiple Myeloma in Non-transplant Candidates: An Entirely Non-intravenous Regimen
Brief Title: Velcade + Cyclophosphamide in Newly Diagnosed Multiple Myeloma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Millennium Pharmaceuticals, Inc. (Industry); Duke Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00038924; Millennium (Other: X05397)
Record Dates: First submitted 2012-11-14; First posted 2012-11-20 (Estimated); Results first posted 2017-05-31 (Actual); Last update posted 2017-05-31 (Actual); Status verified 2017-04

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Bortezomib; Cyclophosphamide; Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Velcade, cyclophosphamide, Revlimid (Experimental): INDUCTION (28-day cycles for 8 cycles):
  * VELCADE 1.3 mg/m2 subcutaneously (SC) days 1, 8 and 15
  * Cyclophosphamide 300 mg/m2 orally (PO) days 1, 8 and 15
  * Dexamethasone 40 mg PO days 1,8 and 15
  MAINTENANCE (28-day alternating cycles until stopped for toxicity, relapse or death):
  * Odd cycles (9, 11, 13, etc.) lenalidomide 10 mg PO days 1-21
  * Even cycles (10, 12, 14, etc.) VELCADE 1.3 mg/m2 SC days 1, 15
  Interventions: Drug: Velcade; Drug: Cyclophosphamide; Drug: Revlimid

INTERVENTIONS:
Drug: Velcade — Bortezomib induction: 1.3 mg/m2, given subcutaneously (SC) on days 1,8 and 15. Up to eight cycles lasting 28 days each will be administered. Patients will not receive any study drugs during the final week of each induction cycle. Bortezomib maintenance (even cycles [10,12,14, etc.]: 1.3 mg/m2, given SC on days 1 and 15. For patients who required VELCADE dose reductions during induction, the last administered mg/m2 dose of VELCADE will be the starting dose for maintenance, given on days 1 and 15. Maintenance cycles will last 28 days and continue indefinitely, until disease progression, lack of tolerability, or death. Patients who cannot tolerate SC VELCADE will be converted to the same dose, given intravenously (IV), per discretion of the treating physician.
  Other Names: bortezomib
Drug: Cyclophosphamide — Cyclophosphamide: 300 mg/m2, given orally on days 1,8 and 15. Up to eight cycles lasting 28 days each will be administered. Patients will not receive any study drugs during the final week of each induction cycle. Patients who cannot swallow cyclophosphamide pills will be converted to the same dose, given intravenously (IV).
Drug: Revlimid — Lenalidomide (odd cycles [9,11,13, etc.]: 10 mg, given orally on days 1-21. Maintenance cycles will last 28 days and continue indefinitely, until disease progression, lack of tolerability, or death. On even cycles, patients will be prescribed enough lenalidomide to take at home, as instructed, for one cycle. This will be prescribed through the mandatory RevlimidREMS® program. If a dose of lenalidomide is missed, it should be taken as soon as possible on the same day. If it is missed for the entire day, it should not be made up.
  Patients who take more than the prescribed dose of lenalidomide should be instructed to seek emergency medical care if needed and contact study staff immediately.
  Other Names: lenalidomide

SUMMARY:
The primary purpose of this study is to estimate the overall response rate (ORR), defined as partial response (PR) or better at any time during induction therapy. The success of the therapy will be determined by ORR with strong consideration given to the secondary endpoints of tolerability, duration of response, and quality of life (QOL).

All patients will be treated with the same experimental regimen. Several novel features are being explored: the substitution of cyclophosphamide for melphalan; once weekly AND subcutaneous bortezomib instead of standard twice weekly, intravenous dosing; and alternating bortezomib and lenalidomide in maintenance.

The investigators hypothesize that this regimen will prove to be tolerable and effective in inducing and maintaining remission in a patient population that is historically very difficult to treat, namely Multiple Myeloma (MM) patients who are too elderly or suffer comorbidities, such as renal insufficiency, that otherwise complicate aggressive therapies like autologous stem-cell transplantation (ASCT). In short, the investigators view this as the "Multiple Myeloma trial for non-trial candidates."

DETAILED DESCRIPTION:
A total of 35 patients will be accrued to this single arm, open label, phase II trial over a period of about 18 months, studying induction chemotherapy with VELCADE, cyclophosphamide and dexamethasone administered on an attenuated dosing schedule to accommodate non-candidates for high-dose chemotherapy with autologous stem cell transplantation - an often frail patient population. Maintenance therapy will follow with alternating lenalidomide and VELCADE. All patients should receive antiviral (zoster) prophylaxis, and peptic ulcer prophylaxis is recommended. Aspirin and/or anticoagulation are left to study physician discretion. All patients will be treated with the same experimental regimen. Several novel features are being explored: the substitution of cyclophosphamide for melphalan; once weekly AND subcutaneous bortezomib instead of standard twice weekly, intravenous dosing; and alternating bortezomib and lenalidomide in maintenance. The overarching aim is to preserve efficacy while minimizing toxicity and inconvenience to this often frail patient population.

ELIGIBILITY:
Inclusion Criteria:

* Voluntary written informed consent before performance of any study-related procedure not part of normal medical care, with the understanding that consent may be withdrawn by the subject at any time without prejudice to future medical care.
* Age ≥18 years at the time of signing the informed consent form.
* Able to adhere to the study visit schedule and other protocol requirements.
* Multiple Myeloma (MM) diagnosed according to the following standard criteria (all three criteria must be met):

  * Monoclonal plasma cells in bone marrow ≥10% and/or presence of biopsy-proven plasmacytoma
  * Laboratory tests meet the levels specified in the protocol
* Measurable disease requiring systemic therapy.
* No prior systemic therapy or radiation therapy active against myeloma lasting more than four weeks duration. Any prior therapy must be completed a minimum of 21 days before starting study drugs. Enrollment of subjects who require radiotherapy (which must be localized in its field size) should be deferred until the radiotherapy is completed and 3 weeks have elapsed since the last date of therapy.
* Karnofsky performance status (KPS) of ≥ 60% at study entry.
* In order to obtain lenalidomide, patients must be registered into the mandatory RevlimidREMS® program during the maintenance phase of therapy, and be willing and able to comply with the requirements of RevlimidREMS®
* Female subjects must be postmenopausal for at least 1 year before the screening visit or surgically sterilized. If females are of childbearing potential, they must adhere to required pregnancy testing; male and female subjects must use specified effective birth control methods.
* Patients should receive concomitant therapy with bisphosphonates, regardless of the presence of bony lesions, although study physicians may use their discretion based on presence of renal insufficiency or other mitigating factors.

Exclusion Criteria:

* Abnormal laboratory tests within the ranges specified in the protocol
* Serum creatinine will not be used to exclude patients. Patients on renal-replacement therapy (e.g., hemodialysis or peritoneal dialysis) will be eligible to participate.
* Light-chain (AL) amyloidosis. Patients with secondary amyloidosis due to MM are eligible.
* ≥ Grade 2 peripheral neuropathy
* Myocardial infarction within 6 months prior to enrollment or has New York Heart Association (NYHA) Class III or IV heart failure, uncontrolled angina, severe uncontrolled ventricular arrhythmias, or electrocardiographic evidence of acute ischemia or active conduction system abnormalities. Prior to study entry, any Electrocardiography (ECG) abnormality at screening must be documented by the investigator as not medically relevant.
* Hypersensitivity to VELCADE, boron, mannitol, or any other component of protocol therapy.
* Female subject is pregnant or lactating. Confirmation that the subject is not pregnant must be established by a negative serum beta-human chorionic gonadotropin (b- hCG) pregnancy test result obtained during screening as specified in section 7.11.
* Female patients who are lactating or have a positive serum pregnancy test during the screening period, or a positive urine pregnancy test on Day 1 before first dose of study drug, if applicable.
* Serious medical or psychiatric illness likely to interfere with participation in this clinical study.
* Diagnosed or treated for another malignancy within 2 years of enrollment, with the exception of complete resection of basal cell carcinoma or squamous cell carcinoma of the skin, an in situ malignancy, or low-risk prostate cancer after curative therapy.
* Participation in clinical trials with other investigational agents not included in this trial, within 14 days of the start of this trial and throughout the duration of this trial.
* Concurrent use of other anti-cancer agents or treatments
* Known HIV positivity
* Known active hepatitis A, B or C

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2012-12-19 (Actual); Primary Completion 2015-12-31 (Actual); Study Completion 2016-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gwynn Long, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 17 subjects consented to the study. 1 subject was a screen failure.
Groups:
- Velcade, Cyclophosphamide, Revlimid: INDUCTION (28-day cycles for 8 cycles):
  * VELCADE 1.3 mg/m2 subcutaneously (SC) days 1, 8 and 15
  * Cyclophosphamide 300 mg/m2 orally (PO) days 1, 8 and 15
  * Dexamethasone 40 mg PO days 1,8 and 15
  MAINTENANCE (28-day alternating cycles until stopped for toxicity, relapse or death):
  * Odd cycles (9, 11, 13, etc.) lenalidomide 10 mg PO days 1-21
  * Even cycles (10, 12, 14, etc.) VELCADE 1.3 mg/m2 SC days 1, 15
  Velcade: Bortezomib induction: 1.3 mg/m2, given subcutaneously (SC) on days 1,8 and 15. Up to eight cycles lasting 28 days each will be administered. Patients will not receive any study drugs during the final week of each induction cycle. Bortezomib maintenance (even cycles [10,12,14, etc.]: 1.3 mg/m2, given SC on days 1 and 15. For patients who required VELCADE dose reductions during induction, the last administered mg/m2 dose of VELCADE will be the starting dose for maintenance, given on days 1 and 15. Maintenance cycles will last 28 days and continue indefinitely, until
Period: Overall Study
Arm/Group | Velcade, Cyclophosphamide, Revlimid
Started | 16
Completed | 14
Not Completed | 2

BASELINE CHARACTERISTICS:
Arm/Group | Velcade, Cyclophosphamide, Revlimid
Number analyzed (Participants) | 14
Age, Continuous [Mean (Standard Deviation); unit: years] | 76.5 (6.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 9

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (ORR) During Induction Therapy
Description: Defined as percentage of patients achieving a partial response or better by International Myeloma Working Group (IMWG) standard criteria:
  IMWG: Complete Response (CR): negative immunofixation on the serum and urine, no soft tissue plasmacytomas and <5% plasma cells in the bone marrow; stringent CR: CR+normal free light chain ratio, no clonal cells in bone marrow by immunohistochemistry or immunofluorescence; Very Good Partial Response: serum and urine M-protein detected by immunofixation but not electrophoresis, >90% in serum M-protein+urine, M-protein level <100 mg/24hour; Partial Response (PR): ≥50% decrease of serum and M-protein, 24 hour urinary M-protein decrease by ≥90% or <200 mg/24hour.
Time Frame: Up to 8 months
Measure: Number; unit: percentage of participants
Arm/Group | Velcade, Cyclophosphamide, Revlimid
Number analyzed (Participants) | 14
percentage of participants | 64

2. Secondary Outcome: Severe Adverse Event Rate
Description: Defined as number of patients experiencing any grade or severe (≥ grade 3 by common toxicity criteria for adverse events (CTCAE) v4.0 criteria) adverse events at any time during the study
Time Frame: Up to 3 years
Measure: Number; unit: percentage of participants
Arm/Group | Velcade, Cyclophosphamide, Revlimid
Number analyzed (Participants) | 14
percentage of participants | 64

3. Secondary Outcome: Maximum Depth of Response During Induction Therapy
Description: Maximum depth of response is defined as: ranging from partial response to complete response by International Myeloma Working Group (IMWG). Described as number of patients achieving each level of response. IMWG: CR: negative immunofixation on the serum and urine, no soft tissue plasmacytomas and <5% plasma cells in the bone marrow; sCR: CR+normal free light chain ratio, no clonal cells in bone marrow by immunohistochemistry or immunofluorescence; VGPR: serum and urine M-protein detected by immunofixation but not electrophoresis, >90% in serum M-protein+urine, M-protein level <100 mg/24hour; PR: ≥50% decrease of serum and M-protein, 24 hour urinary M-protein decrease by ≥90% or <200 mg/24hour. Stable disease mean that the patient has not achieved CR, VGPR, PR or progressive disease.
Time Frame: Up to 8 months
Measure: Number; unit: percentage of participants
Arm/Group | Velcade, Cyclophosphamide, Revlimid
Number analyzed (Participants) | 14
percentage of participants
  Stable Disease | 21
  Partial Response | 7
  Very good partial response (VGPR) | 29
  Complete Response/Stringent complete response | 29
  Progressive Disease/no response | 14

4. Secondary Outcome: Maximum Depth of Response During Maintenance Therapy
Description: Defined as maximum depth of response (ranging from partial response to complete response by International Myeloma Working Group (IMWG) criteria at any point during post-induction maintenance therapy.
  IMWG: Complete Response (CR): negative immunofixation on the serum and urine, no soft tissue plasmacytomas and <5% plasma cells in the bone marrow; stringent CR: CR+normal free light chain ratio, no clonal cells in bone marrow by immunohistochemistry or immunofluorescence; Very Good Partial Response: serum and urine M-protein detected by immunofixation but not electrophoresis, >90% in serum M-protein+urine, M-protein level <100 mg/24hour; Partial Response (PR): ≥50% decrease of serum and M-protein, 24 hour urinary M-protein decrease by ≥90% or <200 mg/24hour. Stable disease mean that the patient has not achieved CR, VGPR, PR or progressive disease.
Time Frame: Up to 3 years
Population: 8 of all subjects reached maintenance and could be analyzed
Measure: Number; unit: percentage of participants
Arm/Group | Velcade, Cyclophosphamide, Revlimid
Number analyzed (Participants) | 8
percentage of participants
  Stable Disease | 13
  Partial Response | 0
  Very good partial response | 50
  Complete Response/Stringent complete response | 38
  Progressive Disease/no response | 0

5. Secondary Outcome: Median Time to Response
Description: Defined as median time to achievement of response (partial remission or better by International Myeloma Working Group standard criteria), in study subjects during 8 months of induction chemotherapy.
Time Frame: Up to 8 months
Measure: Median (Standard Deviation); unit: months
Arm/Group | Velcade, Cyclophosphamide, Revlimid
Number analyzed (Participants) | 14
months | 2 (0.63)

6. Secondary Outcome: Median Duration of Response
Description: Defined as median time elapsed in study subjects between achievement of response and disease progression.
Time Frame: From date of first confirmed response until date of disease progression or up to 3 years
Population: 9 out of all patients achieved response and hence could be analyzed for duration of response
Measure: Median (Standard Deviation); unit: months
Arm/Group | Velcade, Cyclophosphamide, Revlimid
Number analyzed (Participants) | 9
months | 26.2 (0.207)

7. Secondary Outcome: Median Progression-free Survival
Description: Defined as median time elapsed in study subjects between initiation of study therapy and either disease progression or death, regardless of cause of death.
Time Frame: 4 years
Measure: Median (Standard Deviation); unit: months
Arm/Group | Velcade, Cyclophosphamide, Revlimid
Number analyzed (Participants) | 14
months | 24.2 (0.157)

8. Secondary Outcome: Median Overall Survival
Description: Defined as median time elapsed in study subjects between initiation of study therapy and death, regardless of cause.
Time Frame: Up to 3 years
Measure: Median (Standard Deviation); unit: months
Arm/Group | Velcade, Cyclophosphamide, Revlimid
Number analyzed (Participants) | 14
months | 29.7 (0.189)

9. Secondary Outcome: QLQ-C30 Question 29
Description: Measured as mean quality of life in study subjects, quantitatively scored using the standardized and validated European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ). Question 29: how would you rate your overall health during the past week? 7 point scores are standardized to a scale of 0-100, where 100 means highest possible quality.
Time Frame: baseline, 3 months, 5 months
Population: Participants who completed questionnaire.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Velcade, Cyclophosphamide, Revlimid
Number analyzed (Participants) | 10
units on a scale
  Baseline | 58.3 (22.6)
  3 months | 65 (18.9)
  5 months | 68.3 (15.7)
Statistical Analysis 1: Comparison: Velcade, Cyclophosphamide, Revlimid; Test type: Superiority or Other; p = 0.45, paired t-test — Compared baseline to 3 months
Statistical Analysis 2: Comparison: Velcade, Cyclophosphamide, Revlimid; Test type: Superiority or Other; p = 0.19, paired t-test; compares baseline to month 5

10. Secondary Outcome: QLQ-C30 Question 30
Description: Measured as mean quality of life in study subjects, quantitatively scored using the standardized and validated European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ). Question 30: How would you rate your overall quality of life during the past week?
  7 point scores are standardized to a scale of 0-100, where 100 means highest possible quality.
Time Frame: baseline, 3 months, 5 months
Population: Participants who completed questionnaire.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Velcade, Cyclophosphamide, Revlimid
Number analyzed (Participants) | 10
units on a scale
  Baseline | 51.7 (24.1)
  3 months | 66.7 (19.7)
  5 months | 66.7 (12.9)
Statistical Analysis 1: Comparison: Velcade, Cyclophosphamide, Revlimid; Test type: Superiority or Other; p = 0.1, paired t-test — baseline, 3 month
Statistical Analysis 2: Comparison: Velcade, Cyclophosphamide, Revlimid; Test type: Superiority or Other; p = 0.09, paired t-test; baseline, month 5

11. Secondary Outcome: Functionality as Assessed Using the Cancer and Leukemia Group B (CALGB) Geriatric Assessment Tool
Description: Mean functionality in study subjects, quantitatively scored using the standardized and validated Cancer and Leukemia Group B (CALGB) Geriatric Assessment Tool, which comprehensively assesses aspects of a patient's functionality such as symptoms (e.g., pain, anxiety), social support (e.g., someone to turn to for help), and ability to carry out routine activities (e.g., grocery shopping) or physical exertion (e.g., climbing stairs) was assessed at baseline.
  The score is obtained by inserting patient-specific data into the online calculator found at http://www.mycarg.org/Chemo_Toxicity_Calculator, which is based on the risk score described in Hurria A, Togawa K, Mohile SG, et al. Predicting chemotherapy toxicity in older adults with cancer: a prospective multicenter study. J Clin Oncol. 2011;29(25):3457-3465.
  The risk score ranges from 0-19, with 0-5 indicating low risk, 6-9 intermediate risk, and 10-19 high risk for severe (grade >2) toxicity.
Time Frame: baseline
Population: Participants who completed functionality assessment at baseline. Data were incompletely and irregularly collected after baseline so unable to analyze additional time points.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Velcade, Cyclophosphamide, Revlimid
Number analyzed (Participants) | 13
Scores on a scale | 10 (4.5)

12. Secondary Outcome: Risk Score as Assessed Using the Cancer and Leukemia Group B (CALGB) Geriatric Assessment Tool
Description: Calculation of the risk score requires that the patient be assessed with the CALGB Assessment Tool, which has both a patient self-reporting questionnaire and a clinician assessment. Both will be used in this trial, and thus patients will have risk scores based on their own self-assessments and risk scores based on the clinicians' assessment. The risk score ranges from 0-19, with 0-5 indicating low risk, 6-9 intermediate risk, and 10-19 high risk. The distribution of the risk score in this trial will be described by plotting the median of the risk score against time, with patient and clinician assessments overlaid on the same plot.
Time Frame: Day 1
Population: Data for the risk score wasn't recorded correctly, and therefore we were unable to analyze the data.
Arm/Group | Velcade, Cyclophosphamide, Revlimid
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 1st day of drug till 30 days after last dose
Arm/Group | Velcade, Cyclophosphamide, Revlimid
Serious Adverse Events (participants affected / at risk) | 9/14
Other Adverse Events (participants affected / at risk) | 14/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Velcade, Cyclophosphamide, Revlimid (N=14)
Diarrhea (Gastrointestinal disorders) | 1
Infections and infestations - Other, specify (Infections and infestations) | 1
Lung infection (Infections and infestations) | 1
Sepsis (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Fracture (Injury, poisoning and procedural complications) | 1
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 1
Paresthesia (Nervous system disorders) | 1
Delirium (Psychiatric disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Hematoma (Vascular disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Velcade, Cyclophosphamide, Revlimid (N=14)
Anemia (Blood and lymphatic system disorders) | 7 (19)
Cardiac disorders - Other, specify (Cardiac disorders) | 2 (2)
Chest pain - cardiac (Cardiac disorders) | 1 (1)
Ear and labyrinth disorders - Other, specify (Ear and labyrinth disorders) | 1 (1)
Hearing impaired (Ear and labyrinth disorders) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 2 (4)
Blurred vision (Eye disorders) | 2 (3)
Conjunctivitis (Eye disorders) | 1 (1)
Eye disorders - Other, specify (Eye disorders) | 1 (1)
Eye pain (Eye disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (5)
Constipation (Gastrointestinal disorders) | 4 (12)
Diarrhea (Gastrointestinal disorders) | 8 (20)
Dry mouth (Gastrointestinal disorders) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 2 (3)
Mucositis oral (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 5 (11)
Vomiting (Gastrointestinal disorders) | 5 (11)
Chills (General disorders) | 1 (1)
Edema limbs (General disorders) | 8 (10)
Fatigue (General disorders) | 8 (15)
Fever (General disorders) | 2 (2)
Gait disturbance (General disorders) | 2 (2)
General disorders and administration site conditions - Other, specify (General disorders) | 1 (1)
Injection site reaction (General disorders) | 1 (1)
Malaise (General disorders) | 1 (1)
Pain (General disorders) | 1 (1)
Immune system disorders - Other, specify (Immune system disorders) | 1 (1)
Bronchial infection (Infections and infestations) | 1 (1)
Eye infection (Infections and infestations) | 1 (1)
Infections and infestations - Other, specify (Infections and infestations) | 1 (1)
Lung infection (Infections and infestations) | 1 (1)
Skin infection (Infections and infestations) | 2 (2)
Upper respiratory infection (Infections and infestations) | 3 (3)
Urinary tract infection (Infections and infestations) | 3 (4)
Bruising (Injury, poisoning and procedural complications) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1)
Creatinine increased (Investigations) | 5 (8)
Neutrophil count decreased (Investigations) | 5 (8)
Platelet count decreased (Investigations) | 3 (9)
White blood cell decreased (Investigations) | 1 (2)
Anorexia (Metabolism and nutrition disorders) | 1 (3)
Hyperglycemia (Metabolism and nutrition disorders) | 2 (4)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1)
Hyperuricemia (Metabolism and nutrition disorders) | 1 (2)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (1)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 2 (6)
Hypomagnesemia (Metabolism and nutrition disorders) | 3 (4)
Hyponatremia (Metabolism and nutrition disorders) | 1 (2)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (3)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (7)
Bone pain (Musculoskeletal and connective tissue disorders) | 4 (7)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 3 (4)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (6)
Dizziness (Nervous system disorders) | 5 (7)
Dysgeusia (Nervous system disorders) | 1 (2)
Headache (Nervous system disorders) | 2 (2)
Memory impairment (Nervous system disorders) | 2 (2)
Nervous system disorders - Other, specify (Nervous system disorders) | 1 (1)
Paresthesia (Nervous system disorders) | 1 (3)
Peripheral sensory neuropathy (Nervous system disorders) | 5 (9)
Presyncope (Nervous system disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 2 (2)
Confusion (Psychiatric disorders) | 1 (1)
Depression (Psychiatric disorders) | 3 (3)
Insomnia (Psychiatric disorders) | 4 (8)
Libido decreased (Psychiatric disorders) | 1 (1)
Psychiatric disorders - Other, specify (Psychiatric disorders) | 2 (2)
Hematuria (Renal and urinary disorders) | 1 (1)
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 2 (2)
Urinary frequency (Renal and urinary disorders) | 4 (6)
Urinary incontinence (Renal and urinary disorders) | 3 (4)
Urinary tract pain (Renal and urinary disorders) | 2 (4)
Urinary urgency (Renal and urinary disorders) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 5 (14)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 4 (6)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3 (5)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1)
Bullous dermatitis (Skin and subcutaneous tissue disorders) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 8 (16)
Nail loss (Skin and subcutaneous tissue disorders) | 1 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 3 (4)
Purpura (Skin and subcutaneous tissue disorders) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 (3)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 4 (7)
Hot flashes (Vascular disorders) | 3 (3)
Hypertension (Vascular disorders) | 2 (3)
Vascular disorders - Other, specify (Vascular disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No